CLINICAL TRIAL: NCT06021106
Title: The Effect of Respiratory Exercise Applied to COPD Patients With Virtual Reality Glasses on Dyspnea, Anxiety and Quality of Life
Brief Title: Respiratory Exercise to Copd With Virtual Reality Glasses on Dyspnea, Anxiety and Qualıty of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ArdahanU-Simsekli-DS-01
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Copd; Breathing Exercises
Keywords: anxiety; dyspnea; COPD; virtual reality; breathing exercises; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Dyspnea

STUDY DESIGN:
Intervention Model Description: Pretest posttest single blind parallel group randomized controlled experimental study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were not informed about which group they were in, patients in the experimental and control groups were recruited at different times, and separate consent forms were created for the experimental and control groups. The statistician was not informed about the experimental and control groups, and the experimental and control groups were coded as A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Breathing exercises were applied to the experimental group with virtual reality glasses. Each application consists of 20 minutes. The exercises were performed 3 days a week for eight weeks, a total of 24 sessions.
  Interventions: Other: Breathing exercise application with virtual reality glasses
- Control group (Active Comparator): In the control group, routine treatment and care continued and no additional intervention was made.
  Interventions: Other: routine treatment and care

INTERVENTIONS:
Other: Breathing exercise application with virtual reality glasses — In adapting breathing exercises to virtual reality glasses; The exercise video was first shot by the researcher in front of a green screen. Then, a 3D background design was made by a software developer, a 360-degree printout was taken, and it was converted into a form that can be viewed with glasses. The exercise video is prepared as 20 minutes. Exercises were performed at patients' homes through home visits. A total of 24 sessions of exercises were performed three days a week.
  Arms: Experimental group
Other: routine treatment and care — routine treatment and care
  Arms: Control group

SUMMARY:
It was planned to examine the effects of breathing exercises applied with virtual reality glasses on dyspnea, anxiety and quality of life in COPD patients. The study was planned to be conducted in a single-blind pre-test post-test parallel group randomized controlled experimental design. Hypotheses created for the research; H0a: There is no difference between the dyspnea scores of the experimental group and the control group in the post-test in COPD patients. H0b: There is no difference between the anxiety scores of the experimental group and the control group in the post-test in COPD patients. H0c: There is no difference between the quality of life scores of the experimental group and the control group in the post-test in COPD patients. H1a: There is a difference between the dyspnea scores of the experimental group and the control group in the post-test in COPD patients. H1b: There is a difference between the anxiety scores of the experimental group and the control group in the post-test in COPD patients. H1c: There is a difference in quality of life scores between the experimental group and the control group in the post-test in COPD patients. It is planned to apply breathing exercise through virtual reality glasses for 8 weeks to the experimental group. It is planned that the exercises will be done three times a week in a total of 24 sessions. No intervention will be applied to the control group. It is planned to collect the research data in the pre-test, four weeks after the pre-assessment, and in the post-test (in the eighth week of the study). Inclusion criteria for the study; Being over 18 years old, being GOLD Stage II-III COPD (FEV1/FVC<70%, FEV1<80%), being >24 as a result of the mini mental state assessment test, residing in the city center where the research was conducted. Exclusion criteria; exacerbation of COPD for the last four weeks, pneumonia, use of psychiatric medication.

DETAILED DESCRIPTION:
Breathing exercises are the most important part of pulmonary rehabilitation for COPD patients. It helps patients to increase their lung capacity, allowing them to breathe more easily. At the same time, since the patient can easily do breathing exercises by himself, it is also beneficial to provide disease control and self-management. Although breathing exercises are simple and easy to apply, difficulties in the disease process can prevent the individual from doing this. For this reason, there is a need for applications that will attract the attention and interest of patients or direct them, but that will not create commitment to the hospital. In this sense, it has been reported that breathing exercises to be applied through virtual reality glasses will attract the attention and interest of the patient, increase their motivation and make breathing exercises more regular. Therefore, this study was planned to determine the effect of breathing exercises applied with virtual reality glasses on dyspnea, anxiety and quality of life in COPD patients. Material and Method: The study was conducted in a single-blind pre-test post-test parallel group randomized controlled experimental design. The sample size of the study was determined as a result of the power analysis made by taking FEV1% in a study, and considering the losses, it was planned to form the sample of the study of 48 patients, 24 in the experimental and 24 in the control group. In the study, block randomization was chosen to reduce selection bias and distribute patients equally to groups. Patients who accept to participate in the study who meet the inclusion criteria will be pre-tested and assigned to the groups. Since the intervention will be applied in the research, investigator blinding will not be possible, and it is planned to blind the participants, whose consent forms have been prepared separately for the patients in the experimental and control groups. Statistician will be blinded. COPD Patient Identification Form, Pulmonary Function Test Evaluation Form, COPD Evaluation Test (CAT), Modified Medical Research Council (mMRC) Dyspnea Scale, Hospital Anxiety and Depression Scale (HADS), St George Respiratory Questionnaire and Virtual Reality Experience Evaluation Form. Research data will be collected in the pre-test, the fourth week of the research and the post-test (the eighth week of the research). Breathing exercise will be applied to the experimental group with virtual reality glasses. In adapting breathing exercises to virtual reality glasses; The exercise video was first shot by the researcher in front of a green screen. Then, a 3d background design was made by a software developer and it was transformed into a viewable form with these glasses. The exercise video was prepared as 20 minutes. The exercises will be done in the homes of the patients by making home visits. It is planned that the exercises will be done three times a week in a total of 24 sessions. No intervention will be applied to the control group. It is planned to evaluate the research data with the SPSS 26 package program.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being GOLD Stage II-III COPD (FEV1/FVC<70%, FEV1<80%)
* Being oriented and cooperative
* No communication problem
* Being >24 in mini mental state assessment test
* Voluntarily agreeing to participate in the research
* Residing in the center of Ardahan

Exclusion Criteria:

* Exacerbation of COPD in the last 4 weeks
* pneumonia
* Using psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | pretest, week 4, week 8
  refers to the oxygen saturation in the blood
respiratory rate | pretest, week 4, week 8
  refers to the number of breaths per minute
forced vital capacity (FVC) | pretest, week 4, week 8
  This value is the maximum volume of air that can be removed from the lungs by exhaling forcefully, deeply and rapidly after taking a deep breath.
volume of air exhaled in 1 second of forced expiration (FEV1) | pretest, week 4, week 8
  It is the volume expelled in the first second of forced expiration.
Peak Expiratory Flow Rate (PEF) | pretest, week 4, week 8
  It is measured by the maximum exhalation maneuver following the maximum inspiration.
FEV1/FVC | pretest, week 4, week 8
  It is a parameter used to detect the presence of obstruction.
COPD Evaluation Test (CAT) | pretest, week 4, week 8
  Jones et al. (2009) developed this test is used to evaluate the health status of patients with COPD.
Modifiye Medical Research Council (mMRC) | pretest, week 4, week 8
  The scale developed by Fletcher and later edited by the American Thoracic Society was developed to compare the level of dyspnea between individuals with lung disease and those without. The scale is scored between 0-4. The cut off score is 2. High scores indicate severe dyspnea.

SECONDARY OUTCOMES:
Anxiety | pretest, week 4, week 8
  It is a state of fear and anxiety that occurs due to dyspnea in patients with COPD. In this study, the Hospital Anxiety Scale developed by Zigmond and Snaith in 1983 will be used.The scale is scored in a four-likert type. The cutoff score is 10-11. A score above this score means an increased risk in terms of anxiety.
St George's Respiratory Questionnaire (SGRQ) | pretest, week 4, week 8
  It was developed by Jones et al. in 1991 to measure the health-related quality of life of patients with COPD, and its Turkish validity and reliability were performed by Polatlı in 2013. The lowest 0 and the highest 100 points can be obtained. An increase in score indicates worsening of the disease.
Virtual Reality Experience Evaluation Form | pretest, week 4, week 8
  This form was created by scanning the literature in order to evaluate the patient's satisfaction with the breathing exercise with virtual reality glasses applied to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap TAN, Prof. dr., Study Director — Ataturk University
Locations (1):
- Ardahan University, Ardahan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Jang MH, Shin MJ, Shin YB. Pulmonary and Physical Rehabilitation in Critically Ill Patients. Acute Crit Care. 2019 Feb;34(1):1-13. doi: 10.4266/acc.2019.00444. Epub 2019 Feb 28. PMID 31723900
- [Background] Lu Y, Li P, Li N, Wang Z, Li J, Liu X, Wu W. Effects of Home-Based Breathing Exercises in Subjects With COPD. Respir Care. 2020 Mar;65(3):377-387. doi: 10.4187/respcare.07121. Epub 2019 Nov 12. PMID 31719191
- [Background] Marotta N, Demeco A, Moggio L, Marinaro C, Pino I, Barletta M, Petraroli A, Pepe D, Lavano F, Ammendolia A. Comparative effectiveness of breathing exercises in patients with chronic obstructive pulmonary disease. Complement Ther Clin Pract. 2020 Nov;41:101260. doi: 10.1016/j.ctcp.2020.101260. Epub 2020 Nov 17. PMID 33221632
- [Background] Rutkowski S, Szczegielniak J, Szczepanska-Gieracha J. Evaluation of the Efficacy of Immersive Virtual Reality Therapy as a Method Supporting Pulmonary Rehabilitation: A Randomized Controlled Trial. J Clin Med. 2021 Jan 18;10(2):352. doi: 10.3390/jcm10020352. PMID 33477733
- [Background] Condon C, Lam WT, Mosley C, Gough S. A systematic review and meta-analysis of the effectiveness of virtual reality as an exercise intervention for individuals with a respiratory condition. Adv Simul (Lond). 2020 Nov 19;5(1):33. doi: 10.1186/s41077-020-00151-z. PMID 33292807
- [Background] Kanik EA, Taşdelen B, Erdoǧan S. Klinik denemelerde randomizasyon. Marmara Med J. 2011;24(3):149-55. doi: 10.5472/MMJ.2011.01981.1
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415
- [Background] Yorgancioglu A, Polatli M, Aydemir O, Yilmaz Demirci N, Kirkil G, Nayci Atis S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Reliability and validity of Turkish version of COPD assessment test]. Tuberk Toraks. 2012;60(4):314-20. doi: 10.5578/tt.4321. Turkish. PMID 23289460
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Aydemir Ö, Güvenir T, Küey L, Kültür S. Hastane Anksiyete ve Depresyon Ölçeği Türkçe Formunun Geçerlilik ve Güvenilirlik Çalışması. Türk Psikiyatr Derg. 1997;8(4):280-7.
- [Background] Polatli M, Yorgancioglu A, Aydemir O, Yilmaz Demirci N, Kirkil G, Atis Nayci S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Validity and reliability of Turkish version of St. George's respiratory questionnaire]. Tuberk Toraks. 2013;61(2):81-7. doi: 10.5578/tt.5404. Turkish. PMID 23875584
- [Background] Moorhouse N, Jung T, Shi X, Amin F, Newsham J, McCall S. Pulmonary Rehabilitation in Virtual Reality for COPD Patients. 2019;277-90.
- [Background] Garvey C, Bayles MP, Hamm LF, Hill K, Holland A, Limberg TM, Spruit MA. Pulmonary Rehabilitation Exercise Prescription in Chronic Obstructive Pulmonary Disease: Review of Selected Guidelines: AN OFFICIAL STATEMENT FROM THE AMERICAN ASSOCIATION OF CARDIOVASCULAR AND PULMONARY REHABILITATION. J Cardiopulm Rehabil Prev. 2016 Mar-Apr;36(2):75-83. doi: 10.1097/HCR.0000000000000171. PMID 26906147
- [Background] Gloeckl R, Marinov B, Pitta F. Practical recommendations for exercise training in patients with COPD. Eur Respir Rev. 2013 Jun 1;22(128):178-86. doi: 10.1183/09059180.00000513. PMID 23728873
- [Background] Mayer AF, Karloh M, Dos Santos K, de Araujo CLP, Gulart AA. Effects of acute use of pursed-lips breathing during exercise in patients with COPD: a systematic review and meta-analysis. Physiotherapy. 2018 Mar;104(1):9-17. doi: 10.1016/j.physio.2017.08.007. Epub 2017 Aug 31. PMID 28969859
- [Background] Sumedi ., Philip K, Hafizurrachman M. The effect of Pursed Lips Breathing Exercises on the Oxygen Saturation Levels of Patients with Chronic Obstructive Pulmonary Disease in Persahabatan Hospital, Jakarta. KnE Life Sci. 2021;2021:35-64.